CLINICAL TRIAL: NCT04693689
Title: Novelty, Conformity and Trust in Vaccines
Brief Title: Novelty, Conformity and Trust in COVID-19 Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Ho Teck Hua, Director, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SG-Trust in Vaccines
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Trust
Keywords: COVID-19; Coronavirus; Vaccine; Trust; RNA; Global survey
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — mRNA Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Conventional vaccine, 0% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive a conventional vaccine if its current adoption rate in the country is 0%.
  Interventions: Other: Conventional vaccine; Other: 0% adoption rate
- Conventional vaccine, 20% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive a conventional vaccine if its current adoption rate in the country is 20%.
  Interventions: Other: 20% adoption rate; Other: Conventional vaccine
- Conventional vaccine, 40% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive a conventional vaccine if its current adoption rate in the country is 40%.
  Interventions: Other: 40% adoption rate; Other: Conventional vaccine
- Conventional vaccine, 60% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive a conventional vaccine if its current adoption rate in the country is 60%.
  Interventions: Other: 60% adoption rate; Other: Conventional vaccine
- Conventional vaccine, 80% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive a conventional vaccine if its current adoption rate in the country is 80%.
  Interventions: Other: 80% adoption rate; Other: Conventional vaccine
- RNA vaccine, 0% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive an RNA vaccine if its current adoption rate in the country is 0%.
  Interventions: Other: RNA vaccine; Other: 0% adoption rate
- RNA vaccine, 20% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive an RNA vaccine if its current adoption rate in the country is 20%.
  Interventions: Other: RNA vaccine; Other: 20% adoption rate
- RNA vaccine, 40% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive an RNA vaccine if its current adoption rate in the country is 40%.
  Interventions: Other: RNA vaccine; Other: 40% adoption rate
- RNA vaccine, 60% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive an RNA vaccine if its current adoption rate in the country is 60%.
  Interventions: Other: RNA vaccine; Other: 60% adoption rate
- RNA vaccine, 80% adoption rate (Experimental): Our survey follows a 2 x 5 between-subjects design. The two dimensions we vary are vaccine technology (conventional vs. RNA) and the hypothetical adoption rate of the new vaccine in the country (0%, 20%, 40%, 60%, 80%). We elicit subjects' willingness to receive the new COVID-19 vaccine given the vaccine technology and a hypothetical adoption rate of the new vaccine.
  In this arm, we elicit subjects' willingness to receive an RNA vaccine if its current adoption rate in the country is 80%.
  Interventions: Other: RNA vaccine; Other: 80% adoption rate

INTERVENTIONS:
Other: RNA vaccine — We elicit subjects' willingness to receive RNA COVID-19 vaccine
  Arms: RNA vaccine, 0% adoption rate; RNA vaccine, 20% adoption rate; RNA vaccine, 40% adoption rate; RNA vaccine, 60% adoption rate; RNA vaccine, 80% adoption rate
Other: 20% adoption rate — We elicit subjects' willingness to receive the new vaccine if 20% of the country's population has received it
  Arms: Conventional vaccine, 20% adoption rate; RNA vaccine, 20% adoption rate
Other: 40% adoption rate — We elicit subjects' willingness to receive the new vaccine if 40% of the country's population has received it
  Arms: Conventional vaccine, 40% adoption rate; RNA vaccine, 40% adoption rate
Other: 60% adoption rate — We elicit subjects' willingness to receive the new vaccine if 60% of the country's population has received it
  Arms: Conventional vaccine, 60% adoption rate; RNA vaccine, 60% adoption rate
Other: 80% adoption rate — We elicit subjects' willingness to receive the new vaccine if 80% of the country's population has received it
  Arms: Conventional vaccine, 80% adoption rate; RNA vaccine, 80% adoption rate
Other: Conventional vaccine — We elicit subjects' willingness to receive conventional COVID-19 vaccine
  Arms: Conventional vaccine, 0% adoption rate; Conventional vaccine, 20% adoption rate; Conventional vaccine, 40% adoption rate; Conventional vaccine, 60% adoption rate; Conventional vaccine, 80% adoption rate
Other: 0% adoption rate — We elicit subjects' willingness to receive the new vaccine if 0% of the country's population has received it
  Arms: Conventional vaccine, 0% adoption rate; RNA vaccine, 0% adoption rate

SUMMARY:
Despite their established benefits as public measures, vaccines continue to be treated with suspicion by many people, in the US and other parts of the world (Larson et al. 2014; Olive et al. 2018; Lazarus et al. 2020). Since the success of vaccines depends on their high uptake level (Anderson and May, 1985; Fine et al. 2011; Fontanet and Cauchemez, 2020), identifying factors that influence low trust and decision-making in relation to vaccines is essential in order to combat diseases such as the novel Coronavirus (COVID-19).

The investigators study factors that could potentially influence public's trust in COVID-19 vaccines through a large-scale online field experiment. The investigators conduct an online survey of 32,400 subjects in nine countries (USA, Brazil, Mexico, China, India, Indonesia, Russia, Germany, and UK).

The investigators study how willingness to receive the COVID-19 vaccine is affected by (1) the "novelty" of the vaccine technology (conventional vs. RNA vaccines), and (2) the adoption rate of the new vaccine in the country. That is - the impact of controversial science and the force of conformity on the rates of adoption. The latter will also allow us to calculate the "tipping point" adoption rate for each country that will allow the country to achieve herd immunity from COVID-19.

The investigators have four hypotheses, below.

H1 (Conformity): People are more willing to receive a vaccine as the cumulative adoption rate in their community increases.

H2 (Novelty): People are less willing to get a COVID-19 vaccine that uses the new RNA technology, compared to a conventional vaccine

H3 (Interaction between H1 and H2): As the cumulative adoption rate in a community increases, the difference between people's willingness to adopt conventional rather than RNA vaccines decreases.

H4 (Tipping Point): Each country will have a different "tipping point". This is the cumulative adoption rate after which unvaccinated people are significantly more willing to get the vaccine. Countries that have a higher "honesty index" will have the tipping point appear at a lower cumulative adoption rate.

Please note that this study is not a clinical trial. This study is a randomized controlled trial in the form of an online survey.

DETAILED DESCRIPTION:
The investigators study the role of trust in COVID-19 vaccine through a global survey. Specifically, the investigators vary (1) the degree of vaccine innovation and (2) the adoption rate of the vaccine to test if these factors influence the individuals' willingness to receive the vaccine.

An online survey is conducted across 9 countries with 3,600 subjects per country. About 15 questions will be asked for each subject and the survey is expected to take about 10-15 minutes to complete.

The 9 countries are USA, Brazil, Mexico, China, India, Indonesia, Russia, Germany and the UK. The three most populous countries from three major continents (Americas, Asia and Europe) are chosen. The target subjects are healthy adults over 18 years of age.

The survey instrument will consist of two parts. In the first part, the survey will ask 10 questions regarding their demographics and the general perception on the safety, effectiveness, and importance of vaccines. This part of the survey allows us to explore the relationship between the individual factors (such as age, gender or income status) and trust in COVID-19 vaccine, as well as to normalize the attitude towards COVID-19 vaccines over the overall vaccine-related confidence.

The 3 key questions of interest are:

"Suppose that a conventional vaccine for COVID-19 receives approval for human use and is available for the public.

A3. How much do you think the government should subsidize the conventional COVID-19 vaccine? [10%, 25%, 50%, 75%, 100%]

A4. If the conventional COVID-19 vaccine were provided to you for free, how likely are you to accept the vaccination? [Very likely, somewhat likely, neither likely nor unlikely, somewhat unlikely, very unlikely]

A5. Suppose the conventional COVID-19 vaccine is endorsed by your Government, free, but no one in your country has received the vaccine. How likely would you be willing to be vaccinated with this new vaccine? [Very likely, somewhat likely, neither likely nor unlikely, somewhat unlikely, very unlikely]"

The investigators manipulate two dimensions of information between the subjects. The two dimensions are:

* 2 vaccine types: 50% of subjects will be asked for "conventional vaccine"; 50% of subjects will be asked for "RNA vaccine"
* 5 different levels of adoption rate in the country: 0% (i.e., no one in your country has received the vaccine), 20%, 40%, 60%, and 80%

Within each country, there will be 2 (vaccine type) x 5 (different adoption rates) = 10 between-subject treatments.

In the second part of the survey, the investigators ask participants to complete a simple economic dice-rolling task, and predict outcomes of the same task in their own country. The investigators will study how individual performance in these tasks correlate with their trust in COVID-19 vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over 18 years old

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35180 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Willingness to receive COVID-19 vaccine | During the 15-minute survey
  Subjects' response to the question: "If the conventional COVID-19 vaccine were provided to you for free, how likely are you to accept the vaccination?" on a Likert scale from 1 (very unlikely) to 5 (very likely).
Belief in how much COVID-19 vaccine should be subsidized by the government | During the 15-minute survey
  Subjects' response to the question: "How much do you think the government should subsidize the conventional COVID-19 vaccine?" There are 5 answer options: 0%, 25%, 50%, 75%, 100%.

SECONDARY OUTCOMES:
Belief in importance of vaccinating children | During the 15-minute survey
  Subjects' response to the question: "To what extent do you agree or disagree with the following statement: It is important for children to be vaccinated" on a Likert scale from 1 (strongly disagree) to 5 (strongly agree)
Belief in safety of vaccines | During the 15-minute survey
  Subjects' response to the question: "To what extent do you agree or disagree with the following statement: Vaccines are safe" on a Likert scale from 1 (strongly disagree) to 5 (strongly agree)
Belief in effectiveness of vaccines | During the 15-minute survey
  Subjects' response to the question: "To what extent do you agree or disagree with the following statement: Vaccines are effective" on a Likert scale from 1 (strongly disagree) to 5 (strongly agree)
Dishonesty index | During the 15-minute survey
  We ask each subject to report the outcome of a dice roll (which investigators do not observe), where the subject receives a higher pay for reporting a higher roll. We use the average reported dice roll in a group as a measure of the group's dishonesty. A higher number indicates higher degree of dishonesty. If everyone was honest, the average number should be 3.5.

CONTACTS AND LOCATIONS:
Overall Officials: Teck Ho, Principal Investigator — National University of Singapore
Locations (1):
- SurveyMonkey, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will not be storing or sharing any personal identifiers. All individual level data will be anonymized, and only anonymized data will be shared with other researchers, upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After completion of all analyses. It will be made available in the supporting documentation.
Access Criteria: It will be made available in the supporting documentation.

REFERENCES:
- [Background] Anderson RM, May RM. Vaccination and herd immunity to infectious diseases. Nature. 1985 Nov 28-Dec 4;318(6044):323-9. doi: 10.1038/318323a0. PMID 3906406
- [Background] Fine P, Eames K, Heymann DL. "Herd immunity": a rough guide. Clin Infect Dis. 2011 Apr 1;52(7):911-6. doi: 10.1093/cid/cir007. PMID 21427399
- [Background] Fontanet A, Cauchemez S. COVID-19 herd immunity: where are we? Nat Rev Immunol. 2020 Oct;20(10):583-584. doi: 10.1038/s41577-020-00451-5. PMID 32908300
- [Background] Larson HJ, Jarrett C, Eckersberger E, Smith DM, Paterson P. Understanding vaccine hesitancy around vaccines and vaccination from a global perspective: a systematic review of published literature, 2007-2012. Vaccine. 2014 Apr 17;32(19):2150-9. doi: 10.1016/j.vaccine.2014.01.081. Epub 2014 Mar 2. PMID 24598724
- [Background] Lazarus JV, Ratzan SC, Palayew A, Gostin LO, Larson HJ, Rabin K, Kimball S, El-Mohandes A. A global survey of potential acceptance of a COVID-19 vaccine. Nat Med. 2021 Feb;27(2):225-228. doi: 10.1038/s41591-020-1124-9. Epub 2020 Oct 20. PMID 33082575
- [Background] Olive JK, Hotez PJ, Damania A, Nolan MS. The state of the antivaccine movement in the United States: A focused examination of nonmedical exemptions in states and counties. PLoS Med. 2018 Jun 12;15(6):e1002578. doi: 10.1371/journal.pmed.1002578. eCollection 2018 Jun. PMID 29894470

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT04693689/SAP_001.pdf